CLINICAL TRIAL: NCT06399679
Title: Rivastigmine to Prevent Recurrence of Antimuscarinic Delirium After Initial Control With Physostigmine (RIVA-AP): a Randomized, Placebo-controlled Trial
Brief Title: Rivastigmine to Prevent Recurrence of Antimuscarinic Delirium
Acronym: RIVA-AP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Academy of Clinical Toxicology (Other)
Responsible Party: Principal Investigator, Kevin Baumgartner, Assistant Professor of Emergency Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202403052
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Anticholinergic Toxicity
MeSH Terms: interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivastigmine (Experimental): Patients in the rivastigmine arm will receive rivastigmine 3mg by mouth once, followed by rivastigmine 1.5mg by mouth every 1 hour as needed for ongoing delirium or agitation (at the discretion of the treating physician), for up to three doses.
  Interventions: Drug: Rivastigmine
- Placebo (Placebo Comparator): Patients in the placebo arm will receive oral placebo by mouth once, followed by oral placebo every 1 hour as needed for ongoing delirium or agitation (at the discretion of the treating physician), for up to three doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivastigmine — Rivastigmine 3mg by mouth once, followed by rivastigmine 1.5mg by mouth every 1 hour as needed for ongoing delirium or agitation (at the discretion of the treating physician), for a maximum of three doses
  Arms: Rivastigmine
Drug: Placebo — Matching oral placebo by mouth once, followed by placebo by mouth every 1 hour as needed for ongoing delirium or agitation (at the discretion of the treating physician), for a maximum of three doses
  Arms: Placebo

SUMMARY:
Antimuscarinic delirium (AMD) is a common and dangerous toxicology condition caused by poisoning by medications and other chemicals that block muscarinic receptors. Physostigmine is effective in reversing AMD but has a short duration of action, and patient commonly experience recurrence of AMD after initial control with physostigmine.

Recent case reports and small observational studies suggest that rivastigmine, which has a longer duration of action than physostigmine, might be useful in the treatment of AMD. In order to investigate the effectiveness of rivastigmine in preventing recurrence of AMD after initial control with physostigmine, the investigators propose a randomized, placebo-controlled clinical trial of rivastigmine for AMD. The investigators hypothesize that patients treated with rivastigmine after initial control of AMD with physostigmine will experience less recurrence of antimuscarinic delirium than those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* 10 years of age or older
* Diagnosis of antimuscarinic delirium by history and physical examination, in the opinion of the treating attending toxicologist.
* Treatment with physostigmine according to the local standard of care is planned or has been administered by the treating attending toxicologist and is acceptable to the patient's primary attending physician and surrogate decision maker.
* Antimuscarinic delirium is reasonably controlled after initial physostigmine treatment, as determined by treating toxicologist on bedside physical examination. (Patients may begin the screening and enrollment process prior to physostigmine administration, but will not undergo final initiation of study treatment until after response to physostigmine has been confirmed).

Exclusion Criteria:

* Age less than 10 years at time of enrollment
* Surrogate decision maker not available to provide informed consent for enrollment.
* Patient is pregnant or a ward of the state.
* Inability to safely tolerate oral medication, in the judgement of the treating attending physician.
* Evidence of significant risk for serious cardiac or neurologic sequelae of antimuscarinic poisoning:

  a. Any known or suspected seizure activity prior to enrollment b. QRS duration >100 milliseconds on EKG at enrollment c. Any ventricular dysrhythmia prior to enrollment d. Respiratory failure of any etiology requiring endotracheal intubation e. Any hypotension at enrollment: i. Adults: systolic blood pressure (SBP) <90 mmHg ii. Children ≥10: systolic blood pressure (SBP) <90 mmHg, as per Pediatric Advanced Life Support (PALS) age-based cutoff for children 10 years of age or older3 f. Any administration of sodium bicarbonate, hypertonic saline, vasopressors, inotropes, antiarrhythmic agents, or intravenous lipid emulsion prior to enrollment.

  g. Unacceptable risk of serious medical sequelae of antimuscarinic poisoning in the judgment of the treating attending toxicologist.
* Evidence of significant risk of adverse effect of AChE-I:

  a.Bradycardia or risk of AChE-I induced bradycardia at enrollment: i. Adults: heart rate (HR) <80 beats per minute ii. Children: heart rate below the median heart rate for age as proposed by Fleming et al.33:

  1. Ages 10-12: HR <84 beats per minute 2. Ages 12-15: HR <78 beats per minute 3. Ages 15-18: HR <73 beats per minute b. Known or suspected seizure disorder. c. History of asthma or COPD or wheezing during index presentation d. Known or suspected physical obstruction of intestinal or urogenital tract i. Ileus and/or urinary retention due to antimuscarinic poisoning do not exclude patients from enrollment.

  e. Known or suspected peptic ulcer disease.
* Any known allergy or intolerance to rivastigmine or other AChEI.
* Failure to achieve reasonable initial control of antimuscarinic delirium after physostigmine administration, as assessed by treating toxicologist on bedside physical examination.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of AMD recurrence | Typically 8-36 hours after randomization
  Incidence of AMD recurrence, as defined by the development of agitation (Richmond Agitation-Sedation Scale of +1 or higher) and delirium (Confusion Assessment Method for the ICU positive) after initial control of AMD with physostigmine.

SECONDARY OUTCOMES:
Duration of agitation and delirium | Typically 8-36 hours after randomization
  Total duration of time during which patient is experiencing agitation and delirium (defined and assessed as above)
Total amount of sedatives administered | Typically 8-36 hours after randomization
  Total amount of sedatives (antipsychotics, benzodiazepines, dexmedetomidine, propofol, fentanyl, ketamine) administered during the study period.
Use of sedative infusions | Typically 8-36 hours after randomization
  Any use of continuous sedative infusion (dexmedetomidine, benzodiazepine, propofol, fentanyl) during the study period.
Use of physical restraints | Typically 8-36 hours after randomization
  Any use of physical restraints during the study period
Disposition | Typically 8-36 hours after randomization
  Disposition to ICU, stepdown/intermediate care unit, or floor level of care
Time to medical clearance | Typically 8-36 hours after randomization
  Time from presentation to medical clearance by the toxicology consult service
Oversedation | Typically 8-36 hours after randomization
  Incidence of oversedation, defined as RASS lower than -2
Intubation | Typically 8-36 hours after randomization
  Incidence of intubation and mechanical ventilation during the study period
Seizure | Typically 8-36 hours after randomization
  Incidence of epileptic seizure during the study period
Gastrointestinal upset | Typically 8-36 hours after randomization
  Incidence of clinically significant gastrointestinal upset during the study period
Bradycardia | Typically 8-36 hours after randomization
  Incidence of any bradycardia (as defined using age-based heart rate cutoffs) during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Baumgartner, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06399679/ICF_000.pdf